CLINICAL TRIAL: NCT01818401
Title: Medico-economic Interest of the Patient Matched Cutting Blocks (Ancillary) MyKnee ® LBS During the Poses of Complete Prosthesis of Knee GMK ®. Multicentric, Prospective, Controlled, Opened, Randomised Study About a Medical Device.
Brief Title: Medico-economic Interest of the Patient Matched Cutting Blocks (Ancillary) MyKnee ® LBS During the Poses of Complete Prosthesis of Knee GMK ®. Multicentric, Prospective, Controlled, Opened, Randomised Study About a Medical Device. (My Knee)
Acronym: MY Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0100
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis
Keywords: Ancillary tailored; medico-economic study,; total knee replacement; primary or secondary osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): The control group will be constituted of patients with the prosthesis GMK ® without the ancillary MyKnee ® LBS.
  Interventions: Device: the prosthesis GMK ® without the ancillary MyKnee ® LBS
- Matched patient (Other): The treated group will consist of patients which the GMK ® prosthesis with ancillary ® MyKnee LBS.
  Interventions: Device: Matched patient cutting blocks MyKnee ® LBS

INTERVENTIONS:
Device: the prosthesis GMK ® without the ancillary MyKnee ® LBS
  Arms: Control group
Device: Matched patient cutting blocks MyKnee ® LBS
  Arms: Matched patient

SUMMARY:
Over 70.000 total knee arthroplasty (TKA) are performed in France every year, with a 10% yearly increase since the early 1990s. The clinical experience shows a strong rate of success on pain relief and on function. Longevity of the implants has been shown to be determined by the biomechanical design of the prosthesis, and by the implantation technique, especially the correct positioning of the bone cuts during the surgery. To improve the precision of these cuts, the patient matched cutting blocks developed by Medacta allow to adapt the bone cuts to the patient's anatomy, improving the reliability of this procedure. A reduction of the surgery time lengh and bleeding would be other benefits expected with this type of ancillary. The objective of this trial is to study the reliability of patient matched cutting blocks for total knee arthroplasty, by both clinical and radiological assessment, the effect on morbidity reduction during and after the procedure and also the benefit it could bring on an economic point of view.

ELIGIBILITY:
Inclusion Criteria:

all patients requiring a total knee arthroplasty line: primary or secondary osteoarthritis advanced beyond medical treatment.

Exclusion Criteria:

distorded axes or laxity requiring the establishment of constrained prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
compare the functionality of the knee after installation of a total knee replacement between the 2 groups | 2 years after
  The evaluation will use a specific score for total knee arthroplasty: Part of the Knee Society function score (KSS) measured at 1 year after surgery.

SECONDARY OUTCOMES:
to assess knee function by autoquestionnaire KOOS, the KSS knee score, operative time, procedure bleeding, reliability of the ancillary | 2 years after
medico-economic evaluation type "Cost minimization" | 2 years after
  * Compare the costs of implementing the two strategies (A and B) taking into account the resources consumed (operative time, anesthetic drugs, blood bags ...).
  * Determine the least costly therapeutic intervention and medico-economic impact in the current system of financing of hospital expenditure.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nantes, Nantes, France